CLINICAL TRIAL: NCT03768479
Title: The Value of 18F-FES-PET/CT in Predicting the Efficacy of Fulvestrant as First-line Treatment in Postmenopausal Patients With Hormone Receptor-positive Advanced Breast Cancer - a Multicenter Prospective Study
Brief Title: The Value of 18F-FES-PET/CT in Predicting Fulvestrant Efficacy in Breast Cancer
Acronym: PET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XJTU1AF-CRF-2016-020
Record Dates: First submitted 2018-11-26; First posted 2018-12-07 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-06

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FES-Fulvestrant (Experimental): Patients with ER positive breast cancer receive Fulvestrant as the first line treatment enrolled in the study would receive 18F-FES-PET/CT imaging before and after cycle 1 treatment with the first line Fulvestrant.
  Interventions: Device: 18F-FES-PET

INTERVENTIONS:
Device: 18F-FES-PET — 18F-FES-PET/CT imaging before and after cycle 1 treatment with the first line Fulvestrant

SUMMARY:
This study is focused on the value of 18F-FES-PET in predicting the Fulvestrant efficacy in hormone receptor-positive breast cancer. The imaging agent involved in this study is 16α-[18F]-fluoro-17β-estradiol (18F-FES).

DETAILED DESCRIPTION:
This study is an open, multi-center and prospective clinical study, It is the first time investigators are examining this imaging agent in Chinese patients with breast cancer.

The Chinese FDA has approved 18F-FES as an investigational tracer in a selective few research studies. The Chinese FDA has not approved this tracer for any use outside of research. In this research study, the investigators are investigating the use of a PET tracer called 18F-FES in patients with breast cancer.

The purpose is to take images that can measure the amount of a protein called Estrogen Receptor, or 'ER' in breast tumors. The expression level of ER is tightly correlated with the Fulvestrant efficacy in patients with breast cancer. The investigators will take the pictures of the participant's residual tumor lesions using a PET/CT scanner with 18F-FES used as the tracer before and after the first cycle of Fulvestrant treatment. The investigators are trying to clarify the relationship between the clinical Fulvestrant efficacy and the amount change of 18F-FES uptake by breast tumor around the first cycle of Fulvestrant treatment.

This could help them to predict the efficacy of endocrine therapy by monitoring the dynamic levels of ER in advance, and potentially help guide treatment of breast tumors in the future.

18F-FES was initially developed to image the primary breast tumor. In previous studies of 18F-FES conducted in humans, there were no adverse events (there have been no problems). While this is not the first time 18F-FES has been used in humans, it is the first study in which the investigators study its predictive value in the treatment efficacy in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years or older (required for legal consent)
* Have Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Pathologically diagnosed metastatic breast cancer
* Fulvestrant used as the first-line treatment
* Have primary breast tumor that is at least 2 cm in diameter as measured in any dimension on either mammogram, ultrasound, or breast MRI
* Have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

General Exclusion Criteria

* Previously treated metastatic breast cancer
* Concurrent malignancy of any type
* Impaired elimination (as defined as having problems with urination)
* Participation in a research study/studies involving radiation exposure within the past 12 months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, major kidney or liver disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy
* Currently lactating (either breast feeding or breast pumping)

General PET/CT Safety Exclusion Criteria:

* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, steel implants, ferromagnetic objects such as jewelry or metal clips in clothing
* Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest
* Inability to lie comfortably on a bed inside a PET camera for 90 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis)
* Pregnancy: A negative serum pregnancy test is required on the day of the PET procedure for female subjects of child-bearing age.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2017-03-05 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
the change percentage of 18F-FES SUV | At end of cycle 1 of Fulvestrant treatment (each cycle is 28 days)
  The change percentage of 18F-FES standard uptake value (SUV) before and after cycle 1 of Fulvestrant treatment

SECONDARY OUTCOMES:
The correlation between the change percentage of 18F-FES SUV and the clinical efficacy | From the enrollment time to the time of disease progression or 2 years' followup which comes first
  To find the correlation between the change percentage of 18F-FES SUV and the clinical efficacy, and further to determine the cutoff of 18F-FES SUV change percentage that could predict beneficial efficacy of Fulvestrant in breast cancer

OTHER OUTCOMES:
clinical efficacy: RECIST criteria | From the enrollment time to the time of disease progression or 2 years' followup which comes first
  The therapeutic efficacy of Fulvestrant in breast cancer patients, record as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Principal Investigator — First Affiliated Hospital of Xi'an Jiaotong U; Jin Jin, Principal Investigator — First Affiliated Hospital of Xi'an Jiaotong U
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] van Kruchten M, de Vries EG, Glaudemans AW, van Lanschot MC, van Faassen M, Kema IP, Brown M, Schroder CP, de Vries EF, Hospers GA. Measuring residual estrogen receptor availability during fulvestrant therapy in patients with metastatic breast cancer. Cancer Discov. 2015 Jan;5(1):72-81. doi: 10.1158/2159-8290.CD-14-0697. Epub 2014 Nov 7. PMID 25380844